CLINICAL TRIAL: NCT06431789
Title: Prospective Observational Association Between SLCO1B1 Gene Polymorphism and the Anti-factor Xa Activity of Edoxaban in Patients With Moderate to Severe Renal Insufficiency
Status: Recruiting | Type: Observational
Sponsor: Yi Han (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Yi Han, Associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: SLCO1B1
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Gene Polymorphism; Edoxaban; Renal Insufficiency
Keywords: Anti-factor Xa activity; Edoxaban; Moderate to severe renal insufficiency; Solute carrier organic anion transporter family member 1B1
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To provide reference for clinical rational use of edoxaban;
2. Optimize the individualized dosing regimen of edoxaban.

DETAILED DESCRIPTION:
In this study, patients with moderate and severe renal insufficiency receiving edoxaban were selected as research objects. The potential safety of edoxaban in patients with different genotypes was evaluated by detecting the anti-XA factor activity and SLCO1B1 genotyping, so as to optimize the individualized administration regimen of edoxaban.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine clearance of 15-50ml/min was calculated according to the Cockcroft-Gault formula
* Patients who received edoxaban 30mg once daily for more than 5 days for non-valvular atrial fibrillation (CHADS2VAS2 score ≥2) and deep vein thrombosis prevention or treatment
* Patients voluntarily participate and sign informed consent

Exclusion Criteria:

* Age < 18 years old
* Moderate/severe mitral stenosis combined with valvular heart disease, mechanical valve replacement, or rheumatic heart disease
* The patient had used a combination of cyclosporine, erythromycin or ketoconazole or other P-glycoprotein inhibitors within 30 days prior to use or inclusion; Patients were using or had used amiodarone or dronedarone within 30 days prior to inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with edoxaban at the First Affiliated Hospital of Shandong First Medical University (Shandong Qianfo Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Anti-factor Xa activity | six months
  Anti-factor Xa activity

OTHER OUTCOMES:
Safety index:Thrombotic and bleeding events. | six months
  Thrombotic and bleeding events.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Han, doctorate, Principal Investigator — Qianfoshan Hospital
Locations (1):
- First Affiliated Hospital of Shandong First Medical University ( Qianfoshan Hospital of Shandong Province ), Jinan, Shandong, China